CLINICAL TRIAL: NCT02541318
Title: Study of Effects of Dao-In Exercise on the Perimenopausal Women With Sleep Disturbance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MOST 103-2410-H-039-011; Dao-In for Women with Insomnia (Other: Dao-In Exercise Effects on Perimenopausal Women with Insomnia)
Record Dates: First submitted 2015-08-04; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Peri-menopausal Women; Sleep Disturbances; Dao-in Exercise; Body Constitution
Keywords: peri-menopausal women; sleep disturbances; Dao-in exercise; body constitution
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Practice-from Beginning Group (Experimental): The "Practice-from Beginning Group" will practice Duo-in exercise 20 minutes every day for 2 months; while there is no intervention in the "Practice-2 month Later Group". Then, after 2 weeks, the participants of "Practice-from Beginning Group" and "Practice-2 month Later Group" will crossover. The "Practice-from Beginning Group" has no intervention, but the "Practice-2 month Later Group" will practice Duo-in exercise for 2 months.
  Interventions: Behavioral: Duo-in exercise
- Practice-2 month Later Group (Other): The "Practice-from Beginning Group" will practice Duo-in exercise 20 minutes every day for 2 months; while there is no intervention in the "Practice-2 month Later Group". Then, after 2 weeks, the participants of "Practice-from Beginning Group" and "Practice-2 month Later Group" will crossover. The "Practice-from Beginning Group" has no intervention, but the "Practice-2 month Later Group" will practice Duo-in exercise for 2 months.
  Interventions: Behavioral: Duo-in exercise

INTERVENTIONS:
Behavioral: Duo-in exercise — Duo-in exercise was originated from China and with a 5000-years history. Ancient people adopted Duo-in to treat and prevent diseases.

SUMMARY:
Among health problems of peri-menopausal women, sleep disturbances is very common complaint. The aim of this study is to realize the body constitution of the peri-menopausal women with sleep disturbance; and to evaluate the effects of Duo-in practice on this population to see if this intervention can decrease the dosage of hormone replacement therapy.

Quasi-experimental design and convenient sampling are both adopted. Participants will be recruited from China Medical University, Tri-Service General Hospital, Taiwan Society of Health Promotion, and Dr. Chen's Obstetrics and Gynecology Clinic. One hundred of participants who are willing to try Duo-in exercise to improve their sleep quality will be randomly assigned into experiment group and control group. The experiment group will practice Duo-in exercise 20 minutes every day for 2 months; while there is no intervention in the control group. Then, after 2 weeks, the participants of experiment and control group will crossover. The experiment group has no intervention, but the control group will practice Duo-in exercise for 2 months. Chinese version of the Pittsburgh Sleep Quality Index (CPSQI), Body Constitution Questionnaire (BCQ), peri-menopausal disturbance scale, and peri-menopausal fatigue scale will be used in the assessment at each time point. According to previous experience, a total of 70 participants will completed the whole observation course. Generalized estimating equations (GEE) is applied to analyzed the repeated measurement of different time and groups.

This study will provide the evidence for Duo-in exercise as complementary treatment for hormone replacement therapy for peri-menopausal women, and also for integration of Dao-in exercise into mainstream treatment for other patients with sleep disturbance.

ELIGIBILITY:
Inclusion Criteria:

* peri-menopausal women who have sleep disturbances.
* peri-menopausal women who can walk freely and without any disable.

Exclusion Criteria:

* peri-menopausal women who have cancer and other life-threatening diseases.
* peri-menopausal women who have psychological diseases.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) | 2 months after practicing Duo-In
Body Constitution Questionnaire (BCQ) | 2 months after practicing Duo-In

SECONDARY OUTCOMES:
Peri-menopausal disturbance scale | 2 months after practicing Duo-In
Peri-menopausal fatigue scale | 2 months after practicing Duo-In

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chang Su, Ph.D., Principal Investigator — China Medical University, China
Locations (4):
- Taiwan (4):
  - Dr. Chen's Obstetrics and Gynecology Clinic, Hsinchu, Taiwan
  - Taiwan Society of Health Promotion-Taichung Branch, Taichung, Taiwan
  - China Medical Universuty, Taichung, Taiwan
  - Taiwan Society of Health Promotion-Taipei Branch, Taipei, Taiwan